CLINICAL TRIAL: NCT04328376
Title: Measurement of the Electromechanical Window to Improve the Diagnosis of Congenital Long QT Syndrome
Acronym: FEMQT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2019/35
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Long QT Syndrome
Keywords: Long QT syndrome; Electromechanical window; Phonocardiography
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective FEMQT Group (Experimental): Propositus patients with genetically proven LQTS and their relatives
  Interventions: Diagnostic Test: ECG coupled to phonocardiography

INTERVENTIONS:
Diagnostic Test: ECG coupled to phonocardiography — A standard ECG is recorded along with a phonocardiographic recording. The phonocardiographic recording is obtained by using a specific electronic stethoscope plugged into the auxiliary port of the ECG machine. The recording takes less than 30 seconds. The two recording methods are concomitant.
  QT interval is measured on the ECG recording, EMW is measured with ECG coupled to phonocardiography.

SUMMARY:
The goal of this research is to prospectively evaluate the performance of the electromechanical window according to a phonographic method, as a mean of diagnosis of long QT syndrome, and to compare its performance with routine tests used.

DETAILED DESCRIPTION:
Familial long QT syndrome (LQTS) is a hereditary cardiac disorder in which most affected family members have delayed ventricular repolarization manifest on the electrocardiogram (ECG) as QT prolongation. This disease is associated with an increased propensity to palpitations, syncope, polymorphous ventricular tachycardia and sudden arrhythmic death. The diagnosis relies mostly on resting ECG findings and on genetic testing. In clinical practice however, this diagnosis is complicated by 2 main reasons: 1) a significant overlap in ECG findings between healthy and diseased individuals and 2) a frequent identification of genetic variants of unknown significance. Recent studies have suggested that echocardiographic measurement of the electromechanical window (EMW - the delay between the end of mechanical contraction and electrical activation of the heart) has better performance in the diagnosis of LQTS. The echocardiographic technique is however too complicated for routine clinical use. Preliminary work conducted at the University Hospital of Bordeaux and at the University Hospital of Reunion Island has demonstrated that a phonocardiographic approach leads to similar results with an improved feasibility and a good reproducibility.

ELIGIBILITY:
Inclusion Criteria:

* Propositus patients with genetically proven LQTS and their relatives,
* Patients of both sexes aged 12 and over,
* Free, informed and written consent of the patient and the two holders of parental authority for minors.

Exclusion Criteria:

* Inability to consent,
* Person deprived of liberty by judicial or administrative decision,
* Majors subject to a legal protection measure,
* Person participating in another research including an exclusion period still in progress,
* Severely impaired physical and / or psychological health, which, according to the investigator, may affect the participant's compliance with the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Negative predictive value (NPV) obtained by the two methods of diagnosis | Day 1
  The NPV is measured in percentage. The NPV of LQTS diagnosis obtained by phonocardiographic method (measurement of the EMW) and the NPV obtained by standard ECG method (QT measurement prolongation) will be compared.

SECONDARY OUTCOMES:
Values of sensitivity obtained by the two methods of diagnosis | Day 1
  Value of sensitivity is measured in percentage. The values of sensitivity of EMW and standard ECG will be compared.
Values of specificity obtained by the two methods of diagnosis | Day 1
  Value of specificity is measured in percentage. The values of specificity of EMW and standard ECG will be compared.
Positive predictive values obtained by the two methods of diagnosis | Day 1
  Positive predictive value is measured in percentage. Positive predictive values of EMW and standard ECG will be compared.
Area Under the Curves (AUC) obtained by the two methods of diagnosis | Day 1
  The AUC obtained by Receiver Operating Characteristic (ROC) analyses is measured by a value between 0 and 1.
  The AUC obtained by ROC of EMW and standard ECG will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Josselin DUCHATEAU, MD, Principal Investigator — University Hospital, Bordeaux
Locations (4):
- France (4):
  - Nantes University Hospital, Nantes
  - Bordeaux University Hospital, Pessac
  - La Réunion University Hospital, Saint-Pierre
  - Toulouse University Hospital, Toulouse